CLINICAL TRIAL: NCT06779721
Title: Sestrin-2 Levels and Insulin Resistance in Childhood Obesity
Brief Title: Sestrin-2 Levels and Insulin Resistance
Status: Completed | Type: Observational
Sponsor: Kayseri City Hospital (Other Government)
Responsible Party: Principal Investigator, Pembe Soylu Ustkoyuncu, Principal Investigator, Kayseri City Hospital
Other Study IDs: 425/2021
Record Dates: First submitted 2025-01-13; First posted 2025-01-16 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Obese Adolescents
Keywords: Antioxidant; childhood obesity; insulin resistance; sestrin-2; oxidative stress
MeSH Terms: conditions — Pediatric Obesity; Insulin Resistance | interventions — Sesn2 protein, rat

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

INTERVENTIONS:
Other: Sestrin-2 — Sestrin-2 levels were studied in three different groups

SUMMARY:
The aim of this study is to evaluate sestrin-2 levels in children with obesity

ELIGIBILITY:
Inclusion Criteria:

Obese adolescents Body mass index above the 95th percentile BMI Z-score above 2

Exclusion Criteria:

Primary hyperlipidemia Primary liver disease Hypothyroidism Diabetes

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Obese and healthy adolescents who admitted to Kayseri City Hospital
Sampling Method: Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2021-06-20 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of sestrin-2 levels in obese and healthy participants | From enrollment to the end of 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Kayseri City Hospital, Kayseri, Turkey (Türkiye)

REFERENCES:
- [Derived] Soylu Ustkoyuncu P, Kocer D. Sestrin-2 levels and insulin resistance in childhood obesity. J Investig Med. 2025 Jul 7:10815589251359311. doi: 10.1177/10815589251359311. Online ahead of print. PMID 40621934